CLINICAL TRIAL: NCT06286462
Title: Implementing and Evaluating the Cancer Tracking System (CATSystem): A Systems Level Intervention to Improve Cervical Cancer Screening, Treatment Referral and Follow up in Kenya
Brief Title: Evaluation of the Cancer Tracking System (CATSystem)
Acronym: CATSystem
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Global Health Innovations (Other); DARTNet Institute (Other Government); San Diego State University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01CA278617 (NIH)
Record Dates: First submitted 2024-02-06; First posted 2024-02-29 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer
Keywords: cervical cancer screening; treatment of precancerous lesions; treatment of invasive cervical cancer; referral and retention; system level intervention; eHealth intervention; Kenya
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Matched, cluster randomized controlled design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CATSystem Intervention (Experimental): Participants enrolled at intervention sites will receive CATSytem-supported cervical cancer screening and treatment services. Interventions received will include: text messages to patients and algorithm-driven alerts to providers when guideline-adherent cervical cancer screening and treatment services are required including: initial and follow up cervical cancer screening, on site treatment, and referral tracking.
  Interventions: Other: Cancer Tracking System (CATSystem)
- Standard of care (No Intervention): Participants enrolled at control sites will receive standard of care PMTCT services, with no CATSystem tracking or follow up

INTERVENTIONS:
Other: Cancer Tracking System (CATSystem) — The CATSystem provider dashboard highlights patients with overdue services or those in need of outreach and sends automated, customized texts to support screening and treatment follow-up per national guidelines. Points of intervention and alerts include: cervical cancer screening and treatment counseling, initial and follow up cervical cancer screening per national guidelines, treatment for precancer and cancer, referral tracking and follow up. In addition, the CATSystem can securely store images of the cervix taken with colposcopes to allow for remote expert consultation if needed to correctly diagnose a patient or can be reviewed at clinical team meetings for input. Primary goals of the CATSystem are to increase rates of guideline-adherent cervical cancer screening/ rescreening and improve guideline-adherent treatment, referral, and follow-up rates of women with positive screens.
  Arms: CATSystem Intervention

SUMMARY:
Cervical cancer contributes to significant preventable mortality in Kenya where less than 20% of women are screened. The Cancer Tracking System (CATSystem) is a web-based, algorithm generated tool to promote guideline adherent cervical cancer screening and retention through treatment. The goal of this project is to rigorously evaluate the efficacy, implementation, and cost-effectiveness of the CATSystem to improve rates of screening, treatment, referral, and follow-up care in a matched, cluster randomized controlled trial in 10 Kenyan government hospitals (5 intervention, 5 standard of care).

DETAILED DESCRIPTION:
To help address system level barriers to cervical cancer screening, treatment, and follow-up in Kenya, investigators worked with end-users (providers and patients) to develop the Cancer Tracking System (CATSystem), a web-based, algorithm generated tool to promote guideline adherent cervical cancer screening and retention through treatment. The goal of this project is to rigorously evaluate the efficacy, implementation, and cost-effectiveness of the CATSystem to improve rates of screening, treatment, referral, and follow-up care in a matched, cluster randomized controlled trial in 10 Kenyan government hospitals (5 intervention, 5 standard of care). Specific aims (SA) of the study are to (1) Implement and evaluate the efficacy of CATSystem to improve guideline adherent cervical cancer screening, treatment, referral and follow up, (2) Assess feasibility and acceptability of implementation of CATSystem in government run facilities using a human centered design approach, and (3) Calculate the costs and cost-effectiveness of the CATSystem to increase quality adjusted life years gained. Cervical cancer deaths can be prevented with early detection and treatment. This study will evaluate the public health impact of the CATSystem in improving cervical cancer screening, treatment, referral, follow-up, and the feasibility of scale up to other low resource settings.

ELIGIBILITY:
Inclusion Criteria:

* women above 16 years of age
* access to a cell phone,
* presenting for cervical cancer screening at a study hospital.

Exclusion Criteria:

* greater than 20 weeks gestation,
* incarcerated patients,
* women who study staff feel are unable to provide written informed consent due to impaired capacity.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 6600 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Guideline adherent treatment for a positive screen | 0-12 months [from screening result to treatment completion]
  Provide guideline adherent treatment and rescreening for the range of possible positive screen results: cervicitis, precancerous lesions (mild, moderate, severe), invasive cervical cancer. Participants who receive the guideline adherent treatment for their positive screen result will be coded as 1 or "yes". Participants who do not receive the guideline adherent treatment for their positive screen will be coded as 0 or "no".
Cost-effectiveness of the CATSystem Intervention on screening and treatment outcomes | Years 2 and 3
  The cost and cost-effectiveness of the CATSystem to improve Quality-Adjusted Life-Years (QALYs).

SECONDARY OUTCOMES:
Cervical cancer screening | 0-24 months
  Compare the number of women screened for cervical cancer pre (12 month retrospective review of screening rates) and throughout the two-year enrollment period at all intervention and control sites.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Finocchario-Kessler, PhD, Principal Investigator — Univer; Natabhona Mabachi, PhD, Principal Investigator — DARTNet Institute
Locations (10):
- Kenya (10):
  - Akala Health Center, Akala
  - Bondo Referral Hospital, Bondo
  - Alupe Sub-County Hospital, Busia
  - Busia County Referral Hospital, Busia
  - Khunyangu Sub-County Hospital, Busia
  - Matayos Health Center, Busia
  - Port Victoria Sub-County Hospital, Busia
  - Nambale Sub-County Hospital, Siaya
  - Yala Sub-County Hospital, Siaya
  - Ukwala Sub-County Hospital, Ukwala

IPD SHARING:
Plan to Share IPD: Yes
Investigators will make data collected for aims 1 & 2 available only upon request from users who meet eligibility. Data from aim 3 includes costing data for PMTCT services. These data will be shared openly at the dissemination meetings planned at the end of the study, which will include county and national health personnel. Furthermore, these data will be placed in a readily accessible public database.
Supporting Information: Study Protocol, SAP
Time Frame: After participant follow up is complete, data are cleaned, and the data set is locked.
Access Criteria: Eligible requesters are those who can show proof of human subject's training and only under a data-sharing agreement that provides for: (1) use of the data only for research purposes, (2) exclusion of any identifying or potentially identifying information in shared analyses, publications, reports, etc., (3) appropriate storage and securing of the data to prevent authorized persons from accessing it, (4) a commitment to destroy or return the data after analyses are completed.